CLINICAL TRIAL: NCT01555814
Title: Optimization of Treatment and Management of Schizophrenia in Europe (OPTIMISE): the Effects of D2 Antagonism on Candidate Endophenotypes
Brief Title: Optimization of Treatment and Management of Schizophrenia in Europe (OPTIMISE): Substudy Site Copenhagen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birte Glenthoj (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Rigshospitalet, Denmark (Other); Institute of Psychiatry, London (Other); UMC Utrecht (Other); Copenhagen Hospital Corporation (Other)
Responsible Party: Sponsor-Investigator, Birte Glenthoj, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-1-2010-142
Record Dates: First submitted 2011-09-19; First posted 2012-03-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: dopamine; first episode; reward; cognition; MRI; fMRI; PPI; P300; P50 gating; endophenotypes
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amisulpride (Experimental): For 4 weeks, all patients will be treated with amisulpride open label.
  Interventions: Drug: Amisulpride

INTERVENTIONS:
Drug: Amisulpride — 4-week open label amisulpride treatment
  Other Names: Solian

SUMMARY:
The investigators want to relate disturbances in first-episode schizophrenic patients in (dopaminergic) D2 receptors, brain structure, brain function, and information processing to each other and to psychopathology. Additionally, the investigators want to examine the influence of D2 receptor blockade on these disturbances. The investigators expect disturbances in the dopaminergic system at baseline to correlate with specific structural and functional changes and with disruption in information processing as measured with psychophysiological and neurocognitive methods - and investigators expect D2 receptor blockade to reverse some of the functional and cognitive impairments. The investigators do not expect any effect of treatment on brain structure.

DETAILED DESCRIPTION:
The study is designed as a 4 week case-control follow-up study of 90 FE pt. with SCZ and 90 controls matched with regard to age, gender, and parental socio-economic status. All subjects will be examined with a diagnostic interview (SCAN, Schedule for Clinical Assessment in Neuropsychiatry), medical and family history, and physical examination before inclusion. At baseline subjects will be examined with single photon emission computed tomography (SPECT), MRI, fMRI, psychophysiology, neurocognition. In addition, they will be screened for drugs, genetic testing, and ECG. Patients will further be examined with clinical validated rating scales to measure psychopathology, subjective well-being, and side-effects. After a period of 4 weeks all assessments are repeated. During that period patients will be treated with amisulpride, while healthy controls will receive no treatment at all. Efficacy of antipsychotic treatment will be evaluated after this initial period of 4 weeks. All subjects will be re-assessed in the same test battery as mentioned above, except for SPECT and fMRI, after a period of 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia, schizophreniform or schizoaffective disorder (DSM-IV)
* Age 18-40 years
* Written informed consent.

Exclusion Criteria:

* A time interval between the onset of positive symptoms (hallucinations and/or delusions) and study entry exceeding two years.
* Prior use of antipsychotic medication longer than an episode of two weeks in the previous year and/or 6 weeks lifetime.
* Intolerance to one of the drugs in this study. Patients who are coercively treated at a psychiatric ward (based on a judicial ruling)
* Patients who are represented by a legal ward or under legal custody
* The presence of one or more of the contraindications against any of the study drugs as mentioned in the SPC texts
* Pregnancy, as determined through a pregnancy test, or lactation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Relationship between specific neuropsychiatric measures and global improvement on PANSS scores | 4 weeks of medical treatment
  Changes in neuropsychiatric measures like (e.g. PPI, P50-suppression, neurocogtion etc.) will be evaluated and related to the primary outcome measure of the main OPTiMiSE study, the PANSS score change from baseline to follow-up.

SECONDARY OUTCOMES:
Effect of antipsychotic medication on the D2 binding potential (SPECT) in antipsychotic naive patients with schizophrenia. | Baseline, 4 weeks
  D2 receptor binding will be evaluated at baseline and after 4 weeks of treatment. This will be related to measures of the human reward system.
Effect of antipsychotic medication on P50-suppression | Baseline, 4 weeks, 6,12,24 months
  Time/dose improvement on P50 suppression after antipsychotic treatment
Effect of antipsychotic medication on the human reward system | Baseline and 4 weeks follow up
  Disturbances in the human reward system in antipsychotic naive patients with schizophrenia will be evaulated using a reward related BOLD fMRI paradigme.
Change in hippocampal and basal ganglia volume from baseline to follow-up. | 4 weeks, 6, 12 and 24 months,
  Hippocampal volume decrease and basal ganglia volume increase is expected longitudinal outcomes.
Change in processing speed over time after antipsychotic treatment. | Baseline, 4 weeks, 6,12,24 months
  Processing speed is expected to improve.
Change in levels of brain perfusion from baseline to follow-up. | Baseline, 4 weeks treatment
  Brain perfusion levels will be measured in brain areas related to the human reward systems.

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthøj, MD, DMSc, Principal Investigator — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup Glostrup, Denmark
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup Glostrup, Denmark, Glostrup Municipality, Denmark

REFERENCES:
- See also: Site home page — http://cnsr.dk
- See also: Site home page — http://www.cinsr.dk